CLINICAL TRIAL: NCT00044538
Title: An Uncontrolled, Phase II Study Evaluating Anti-Tumor Efficacy and Safety of BAY 59-8862 in Patients With Taxane Resistant Non-Small Cell Lung Carcinoma (NSCLC)
Brief Title: Evaluation of BAY 59-8862 in Taxane Resistant Non-Small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10653
Record Dates: First submitted 2002-08-30; First posted 2002-09-04 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Taxane; Lung cancer, non-small cell; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — IDN 5109

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: BAY59-8862 (Cytotoxic Taxane)

INTERVENTIONS:
Drug: BAY59-8862 (Cytotoxic Taxane) — Intravenous dose over 60 minutes every 3 weeks

SUMMARY:
Lung cancer is among the most common cancers in the world and its incidence continues to increase. Chemotherapy for patients with Non-Small Cell Lung Cancer (NSCLC) has been under investigation for several decades and several new drugs with activity in NSCLC have been identified. These include the taxanes, which are among the most commonly used class of chemotherapy agents in clinical oncology today. The usefulness of the taxanes is limited by the development of tumor resistance to these agents. This phase II trial with BAY 59-8862 will be conducted to determine the anti-tumor efficacy of BAY 59-8862 in taxane-resistant NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease as defined by the presence of at least one measurable lesion
* Patients must have received at least 3 weeks of continuous therapy with Taxane - patient must subsequently develop progressive disease either during treatment or within 6 months after treatment
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver and kidney function

Exclusion Criteria:

* Excluded medical conditions like: pre-existing neuropathy, active heart diseases or ischemia, serious infections, HIV infection, chronic hepatitis B or C; brain metastasis, seizures, hypersensitivity to taxanes, organ transplants, some previous cancers
* excluded therapies and medications, previous and concomitant such as: anticancer chemotherapy or immunotherapy during the study or within 4 weeks prior to study entry; more than two prior anticancer chemotherapy regimens; radiotherapy during study or within 4 weeks prior to study entry; bone marrow transplant.
* others: pregnant or breast-feeding patients; both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial; substance abuse, medical, psychological or social conditions that may interfere with the patient's participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2001-12; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (26):
- United States (7):
  - Tucson, Arizona
  - Waterbury, Connecticut
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Buffalo, New York
  - Columbus, Ohio
  - Nashville, Tennessee
- Canada (5):
  - Edmonton, Alberta
  - Hamilton, Ontario
  - Thunder Bay, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Germany (2):
  - Gauting, Bavaria
  - Berlin, State of Berlin
- Israel (3):
  - Kfar Saba
  - Tel Aviv
  - Tel Litwinsky
- Italy (5):
  - Modena
  - Parma
  - Pisa
  - Torino
  - Udine
- Spain (4):
  - Elche, Alicante
  - Barcelona, Barcelona
  - Barakaldo, Bizkaia
  - Madrid, Madrid